CLINICAL TRIAL: NCT06824077
Title: A Randomised, Placebo Controlled Clinical Trial of Dexmedetomidine as Part of a Sleep Promotion Bundle to Improve Sleep in Intensive Care
Brief Title: Reducing Days DELirious With DEXmedetomidine as Part of an Intensive Care Unit Sleep Promotion Bundle
Acronym: DELDEX
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00147451
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Delirium; ICU Hospitalization
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dexmedetomidine will be prepared at a concentration of 4 mcg/ml by diluting 200 mcg/2 ml vials with 48 mL of 0.9% normal saline to a total volume of 50 ml. A maintenance infusion of 0.2-1.2 mcg/kg/hr will be initiated to sustain the sedative effect and promote sleep throughout the trial period. ICU nurses are experienced in titrating dexmedetomidine for both patients on high flow oxygen (optiflow) and intubated patients with delirium as part of routine care.
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Patients randomized to the control group will receive a placebo daily for 2 consecutive nights.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be prepared at a concentration of 4 mcg/ml by diluting 200 mcg/2 ml vials with 48 mL of 0.9% normal saline to a total volume of 50 ml. A maintenance infusion of 0.2-1.2 mcg/kg/hr will be initiated to sustain the sedative effect and promote sleep throughout the trial period. ICU nurses are experienced in titrating dexmedetomidine for both patients on high flow oxygen (Optiflow) and intubated patients with delirium as part of routine care. The ICU bedside nurse will be responsible for using the lowest effective dose to achieve a Richmond Agitation Sedation Scale (RASS) of -2, up to a maximum of 1.2 mcg/kg/hr, while monitoring for adverse events such as bradycardia and hypotension.
  Arms: Intervention
Other: Control (placebo) group — The control group will receive an infusion of 0.9% saline at 5-45 ml/hr titrated to the lowest effective dose to achieve a RASS of -2 for two nights following randomization.
  Arms: Control

SUMMARY:
Patients frequently experience problems with sleep while admitted to the ICU. Good sleep is important in ensuring that your immune system responds properly to infection, for your heart to function optimally, and to support normal brain function such as memory.

To address sleep problems in the ICU, a bundle of interventions to support more normal sleep are provided. These bundles consist of medications such as sedatives and environmental changes such as less frequent times being assessed overnight and noise reduction strategies. Although medications can make patients appear to be sleeping, most medications do not provide patients with restful sleep. More research is needed on medications that better mimick restful sleep. One such medication is dexmedetomidine. When formally measured dexmedetomidine can make sleep appear more like a patient sleeping at home as compared to the hospital.

The purpose of this study is to test whether giving a patient in the intensive care unit dexmedetomidine helps have a more restful sleep and possibly be more alert and/or interactive the next day.

To see if dexmedetomidine improves sleep, the investigators will compare the quality of sleep of two different groups of participants: one group that receives dexmedetomidine at night for 2 nights in a row and another group that does not. How well one sleeps will be measured, in either group, will be assessed by a portable sleep machine that is attached by several stickers.

This study is called a pilot or feasibility study. A pilot study assesses how easy it is to recruit patients, whether the sleep machine is tolerated, and amount of time sleep is measured.

It is anticipated that about 50 people will take part in this study. This study should take approximately 2 years to complete, and the results should be known in about 1-2 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 years old or over admitted to the ICU
* Anticipated to stay in the ICU for another 48 hours after the first sleep recording
* Mechanically ventilated or on high flow oxygen (Optiflow)
* Hemodynamically stable
* Conscious, non-sedated patient with capacity to complete a self-reported sleep assessment*

Exclusion Criteria:

* Contraindication to dexmedetomidine (including but not limited to allergy and bradycardia [heart rate < 50 beats per minute])
* Currently receiving dexmedetomidine or other alpha-2 agonists (e.g., clonidine)
* Patients with structural neurological disease (e.g., stroke or tumor or traumatic brain injury) or degenerative neurologic disease (e.g., Parkinson's disease or dementia) and GCS < 14
* Patients with second- or third-degree heart block (unless pacemaker implanted)
* Patients with clinically significant hepatic or renal disease
* Patients with limitations in therapy or actively being palliated
* Patients with primary psychiatric disorder (e.g., new diagnosis of or uncontrolled schizophrenia, severe depression)
* Patients experiencing substance intoxication or withdrawal (e.g., severely agitated delirium)
* Patients participating in other studies involving the use of pharmacologically active substances
* Treating clinician believes study participation is not in the patient's best interest
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 years
  Rate of recruitment: The investigators will consider the main trial to be feasible if a recruitment rate of at least 1 patient per month per participating site is achieved. The investigators will report recruitment rates with 95% confidence intervals.

SECONDARY OUTCOMES:
Protocol Adherence | 2 years
  Adherence to treatment duration protocol: The investigators will consider the main trial to be feasible if intervention is delivered 90% of scheduled duration (proportion of total hours study drug received during intervention period (20:00 - 06:00). Further, tolerance of Prodigy Sleep Machine will be evaluated for a similar proportion of time successfully worn (recordings that are of sufficient quality to permit analyses between 20:00 - 06:00). The investigators will report proportion of adherence with 95% confidence intervals.

IPD SHARING:
Plan to Share IPD: Undecided